CLINICAL TRIAL: NCT00061074
Title: The Effects of ERT on Appetitive Behavior and Withdrawal in Short-term Smoking Cessation in Postmenopausal Females on Transdermal Nicotine Replacement
Brief Title: Tobacco Cessation in Postmenopausal Women (Part II) - 2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-08075-2; R01DA008075-02 (NIH)
Record Dates: First submitted 2003-05-21; First posted 2003-05-22 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Tobacco Use Disorder
Keywords: Smoking
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Nicotrol

SUMMARY:
The purpose of this study is to evaluate the effects of ERT on appetitive behavior and withdrawal in short-term smoking cessation in postmenopausal females on transdermal nicotine replacement

ELIGIBILITY:
Inclusion Criteria:

(Same as Part I)

Exclusion Criteria:

Same as Part I, with the addition of those who have had a past reaction to transdermal nicotine patch or have active skin diseases will be excluded.

Ages: 40 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 1993-03; Primary Completion 2000-03 (Actual); Study Completion 2000-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Allen, Ph.D., M.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States